CLINICAL TRIAL: NCT00918879
Title: A 24-Week National, Multi-centre, Randomized, Parallel-group, Double-blind, Placebo-controlled, Phase IIIb Study in India to Evaluate the Efficacy and Safety of Saxagliptin in Adult Patients With Type 2 Diabetes Who Have Inadequate Glycaemic Control With Diet and Exercise
Brief Title: Evaluate Saxagliptin in Adult Indian Patients With Type 2 Diabetes Inadequate Glycemic Control
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: AstraZeneca, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D1680C00008
Record Dates: First submitted 2009-06-05; First posted 2009-06-11 (Estimated); Results first posted 2011-09-26 (Estimated); Last update posted 2011-09-26 (Estimated); Status verified 2011-08

CONDITIONS: Type 2 Diabetes
Keywords: DPP-4 inhibitors; HbA1c; Incretins
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — saxagliptin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Saxagliptin
  Interventions: Drug: Saxagliptin
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Saxagliptin — Oral tablet, once daily for 24 weeks
  Other Names: Onglyza
  Arms: 1
Drug: Placebo — Oral tablet, once daily for 24 weeks
  Arms: 2

SUMMARY:
Saxagliptin is a new investigational medication being developed for treatment of type 2 diabetes. This study is designed to evaluate the efficacy and safety in adult Indian patients with inadequate glycaemic control with diet and exercise.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Type 2 diabetes
* Patients should be drug naïve ie, not received medical treatment for diabetes
* HbA1c ≥ 7.2% and ≤10.0% (at enrolment), HbA1c ≥ 7.0% and ≤10.0% (at randomization)

Exclusion Criteria:

* Insulin therapy within one year of enrolment (with the exception of insulin therapy during a hospitalization or use in gestational diabetes)
* Type 1 diabetes,history of ketoacidosis or hyperosmolar non-ketonic koma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2009-05; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Ohman, MD, PhD, Study Director — AstraZeneca, Wilmington, USA; Deborah Price, MSc, Study Chair — AstraZeneca, Wilmington, USA
Locations (9):
- India (9):
  - Research Site, Gujarat, Ahmedabad
  - Research Site, Karnataka, Bangalore
  - Research Site, Tamil Nadu, Chennai
  - Research Site, Tamil Nadu, Coimbatore
  - Research Site, Andhra Pradesh, Hyderabad
  - Research Site, Madhya Pradesh, Indore
  - Research Site, Haryāna, Karnal
  - Research Site, Kerala, Kochi
  - Research Site, Maharashtra, Pune

REFERENCES:
- [Derived] Perl S, Cook W, Wei C, Iqbal N, Hirshberg B. Saxagliptin Efficacy and Safety in Patients With Type 2 Diabetes and Moderate Renal Impairment. Diabetes Ther. 2016 Sep;7(3):527-35. doi: 10.1007/s13300-016-0184-9. Epub 2016 Jul 11. PMID 27402391

RESULTS

PARTICIPANT FLOW:
Groups:
- Saxagliptin 5 mg: Saxagliptin 5 mg tablet, once daily( OD) for 24 weeks
- Placebo: Placebo tablet, once daily( OD) for 24 weeks
Period: Overall Study
Arm/Group | Saxagliptin 5 mg | Placebo
Started | 107 (Randomized and treated) | 106 (Randomized and treated)
Completed | 101 (Completed 24 weeks of treatment) | 100 (Completed 24 weeks of treatment)
Not Completed | 6 | 6
Not completed — Withdrawal by Subject | 4 | 4
Not completed — Lost to Follow-up | 1 | 1
Not completed — Severe non-compliance to protocol | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Saxagliptin 5 mg | Placebo | Total
Number analyzed (Participants) | 107 | 106 | 213
Age Continuous [Mean (Standard Deviation); unit: Years] | 49.07 (8.77) | 48.29 (9.59) | 48.68 (9.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 43 | 93
  Male | 57 | 63 | 120

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline to Week 24 in Glycosylated Haemoglobin A1c (HbA1c)
Description: Adjusted* mean change from baseline in glycosylated haemoglobin A1c (HbA1c) achieved with saxagliptin 5 mg versus placebo at Week 24 (LOCF, Full Analysis set). HbA1c is a continuous measure, the change from baseline for each subject is calculated as the Week 24 values minus the baseline value. HbA1c data were excluded on and after rescue medication.
Time Frame: Baseline , Week 24
Population: Randomized participants who took at least 1 dose of double-blind treatment. To be included in analysis of change from baseline to Wk 24(LOCF) for efficacy, subjects must have had a baseline and at least 1 post-baseline efficacy measurement. If participant received rescue medication, that measurement must have been taken before rescue.
Measure: Mean (Standard Error); unit: percent
Arm/Group | Saxagliptin 5 mg | Placebo
Number analyzed (Participants) | 104 | 105
percent
  Baseline | 8.33 (0.080) | 8.33 (0.072)
  Week 24 | 7.82 (0.116) | 8.28 (0.114)
  Adjusted Change from Baseline to Week 24 | -0.51 (0.098) | -0.05 (0.098)
Statistical Analysis 1: Comparison: Saxagliptin 5 mg vs Placebo; Test type: Superiority or Other; p = 0.0011, ANCOVA; * adjusted for baseline HbA1c; Mean Difference (Net) = -0.46, 95% CI [-0.73 to -0.18], Standard Error of Mean 0.139

2. Secondary Outcome: Absolute Change From Baseline to Week 24 in Fasting Plasma Glucose (FPG)
Description: Adjusted* mean change from baseline in fasting plasma glucose (FPG) achieved with saxagliptin 5 mg versus placebo at Week 24 (LOCF, Full Analysis set). FPG is a continuous measure, the change from baseline for each subject is calculated as the Week 24 values minus the baseline value. FPG data were excluded on and after rescue medication.
Time Frame: Baseline , Week 24
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Saxagliptin 5 mg | Placebo
Number analyzed (Participants) | 106 | 104
mg/dL
  Baseline | 150.77 (3.569) | 151.35 (3.693)
  Week 24 | 140.58 (3.326) | 151.02 (4.833)
  Adjusted Change from Baseline to Week 24 | -10.35 (3.827) | -0.16 (3.863)
Statistical Analysis 1: Comparison: Saxagliptin 5 mg vs Placebo; Test type: Superiority or Other; p = 0.0623, ANCOVA; * Adjusted for baseline FPG; Mean Difference (Net) = -10.19, 95% CI [-20.91 to 0.53], Standard Error of Mean 5.438

3. Secondary Outcome: Absolute Change From Baseline to Week 24 in Fasting Plasma Glucose (FPG)
Description: as for outcome 2
Time Frame: Baseline , Week 24
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Saxagliptin 5 mg | Placebo
Number analyzed (Participants) | 106 | 104
mmol/L
  Baseline | 8.37 (0.198) | 8.40 (0.205)
  Week 24 | 7.80 (0.185) | 8.38 (0.268)
  Adjusted Change from Baseline to Week 24 | -0.58 (0.212) | -0.00 (0.214)
Statistical Analysis 1: Comparison: Saxagliptin 5 mg vs Placebo; Test type: Superiority or Other; p = 0.0623, ANCOVA; * Adjusted for baseline FPG; Mean Difference (Net) = -0.57, 95% CI [-1.17 to 0.02], Standard Error of Mean 0.302

4. Secondary Outcome: Proportion of Patients (Expressed in Percentage of Total Participants) Achieving a Therapeutic Glycemic Response Defined as HbA1c < 7.0% at Week 24
Description: Proportion of participants (expressed in percentage of total participants)achieving HbA1c < 7.0% for saxagliptin versus placebo at Week 24 (LOCF, Full Analysis set). HbA1c data were excluded on and after rescue medication
Time Frame: Baseline , Week 24
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Saxagliptin 5 mg | Placebo
Number analyzed (Participants) | 104 | 105
Percentage of Participants | 22.1 | 13.3
Statistical Analysis 1: Comparison: Saxagliptin 5 mg vs Placebo; Test type: Superiority or Other; Fisher Exact; Mean Difference (Net) = 8.8, 95% CI [-1.7 to 19.3]

ADVERSE EVENTS:
Arm/Group | Saxagliptin 5 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/107 | 0/106
Other Adverse Events (participants affected / at risk) | 9/107 | 10/106
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Saxagliptin 5 mg (N=107) | Placebo (N=106)
Urinary Tract Infection (Infections and infestations) | 9 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No